CLINICAL TRIAL: NCT01642147
Title: Cerebral Hyperemia During Emergence From General Anesthesia for Craniotomy of Patients With Brain Tumor
Brief Title: Cerebral Blood Perfusion Changes After General Anesthesia for Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Yu Yang, Principal Investigator, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY2012-183
Record Dates: First submitted 2012-07-08; First posted 2012-07-17 (Estimated); Results first posted 2013-04-23 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Brain Neoplasms; Surgery; Hyperemia
Keywords: Cerebral blood flow; Transcranial Doppler; Emergence from general anesthesia
MeSH Terms: conditions — Brain Neoplasms; Hyperemia | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients undergoing craniotomy (Experimental): Patients undergoing craniotomy who are scheduled for selective supratentorial tumor removal surgery will be randomly chosen and recruited.
  Transcranial Doppler (TCD) measures,jugular venous bulb catheterization, radial artery catheterization, and tumor removal surgery under general anesthesia will be performed.
  Interventions: Device: Transcranial Doppler (TCD); Procedure: jugular venous bulb catheterization; Procedure: Tumor removal surgery under general anesthesia; Procedure: Radial artery catheterization
- Patients undergoing abdominal surgery (Active Comparator): Randomly chosen patients undergoing selective abdominal surgery. Transcranial Doppler (TCD) measures,radial artery catheterization, and major abdominal surgery under general anesthesia will be performed.
  Interventions: Device: Transcranial Doppler (TCD); Procedure: Radial artery catheterization; Procedure: Abdominal surgery under general anesthesia

INTERVENTIONS:
Device: Transcranial Doppler (TCD) — A 2-MHz Transcranial Doppler probe (MULTI-DOP P2.2C; DWL, Elektronische Systeme GmbH, Germany) will be used to measure both sides of Vmca of both patients undergoing craniotomy and patients undergoing abdominal surgery. The signal will be range-gated to a depth of 45 to 60 mm at temporal bone window to achieve the optimal signal according to standard techniques. The measures will be recorded in the operation room before anesthesia, in the recovery room at extubation, 30, 60, 90, and 120 min after extubation.
  Other Names: TCD
Procedure: jugular venous bulb catheterization — After local anesthesia, a jugular venous bulb catheter(16G, manufactured by Arrow International Inc. USA) will be placed in the dominant side. The proper placement of the tip of the catheter in the jugular bulb will be confirmed later by a postoperative lateral skull X-ray. SjvO2 (blood sample will be drawn slowly at a speed of 2ml per minute) will be measured before anesthesia, at extubation, 30, 60, 90, and 120 min after extubation.
  Other Names: blood oxygen saturation of jugular vein bulb (SjvO2)
  Arms: Patients undergoing craniotomy
Procedure: Tumor removal surgery under general anesthesia — Surgery types include total or subtotal removal of tumors.For all surgical procedures, general anesthesia will be maintained with isoflurane (0.5-1.0 minimal alveolar concentration (MAC) expired), repeated boluses of fentanyl (1~2 µg/kg IV), and continuous vecuronium 50～70 IV. All patients will be mechanical ventilated with oxygen. During anesthesia, blood pressure and heart rate will be kept stable, within ±10% of the preoperative levels. Hematocrit (Hct) will be maintained higher than 30%. After surgery, tracheal extubation will be performed when patients regain full muscle strength, breathe spontaneously with acceptable oxygenation and normocapnia.
  Other Names: craniotomy under general anesthesia
  Arms: Patients undergoing craniotomy
Procedure: Radial artery catheterization — After local anesthesia, an intra-arterial pressure line(I.V. catheter and pressure line kit are both manufactured by Smiths Medical International Ltd. USA) will be inserted in radial artery. Sample blood will be drawn from the line before anesthesia, at tracheal extubation, and 30, 60, 90, 120 min after tracheal extubation.
Procedure: Abdominal surgery under general anesthesia — For all surgical procedures, general anesthesia will be maintained with isoflurane (0.5-1.0 minimal alveolar concentration (MAC) expired), repeated boluses of fentanyl (1~2 µg/kg IV), and continuous vecuronium 50～70 IV. All patients will be mechanical ventilated with oxygen. During anesthesia, blood pressure and heart rate will be kept stable, within ±10% of the preoperative levels. Hematocrit (Hct) will be maintained higher than 30%. After surgery, tracheal extubation will be performed when patients regain full muscle strength, breathe spontaneously with acceptable oxygenation and normocapnia.
  Arms: Patients undergoing abdominal surgery

SUMMARY:
Few studies look into cerebral blood flow (CBF) changes during emergence from general anesthesia for craniotomy. The purpose of this study is to demonstrate CBF changes during emergence from general anesthesia for craniotomy, through monitoring blood oxygen saturation of jugular vein bulb and transcranial Doppler.

DETAILED DESCRIPTION:
30 patients undergoing selective craniotomy (craniotomy group) for supratentorial brain tumor removal and 30 patients undergoing selective abdominal surgery (abdominal surgery group) are planned to be enrolled in the study. Mean blood flow velocity in middle cerebral artery (Vmca), mean arterial pressure (MAP), blood oxygen saturation of jugular vein bulb (SjvO2) (only measured in craniotomy group)and arterial CO2 partial pressure (PaCO2) will be measured before general anesthesia, at tracheal extubation, and 30,60, 90, 120 min after extubation in both groups.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) physical status I or II
* Scheduled for selective supratentorial tumor removal surgery or major abdominal surgery.

Exclusion Criteria:

* Patients with evidence of systemic hypertension, intracranial hypertension, cerebrovascular diseases, other coexisting medical conditions likely to affect cerebral autoregulation.
* Preoperatively planned delayed tracheal extubation.
* Pregnant or nursing women

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Yu Yang, Master, Principal Investigator — Huashan Hospital; Shou-Jing Zhou, Master, Study Chair — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Rasmussen M, Juul N, Christensen SM, Jonsdottir KY, Gyldensted C, Vestergaard-Poulsen P, Cold GE, Ostergaard L. Cerebral blood flow, blood volume, and mean transit time responses to propofol and indomethacin in peritumor and contralateral brain regions: perioperative perfusion-weighted magnetic resonance imaging in patients with brain tumors. Anesthesiology. 2010 Jan;112(1):50-6. doi: 10.1097/ALN.0b013e3181c38bd3. PMID 19952725
- [Background] Randell T, Niskanen M. Management of physiological variables in neuroanaesthesia: maintaining homeostasis during intracranial surgery. Curr Opin Anaesthesiol. 2006 Oct;19(5):492-7. doi: 10.1097/01.aco.0000245273.92163.8e. PMID 16960480
- [Background] Clavier N, Schurando P, Raggueneau JL, Payen DM. Continuous jugular bulb venous oxygen saturation validation and variations during intracranial aneurysm surgery. J Crit Care. 1997 Sep;12(3):112-9. doi: 10.1016/s0883-9441(97)90040-x. PMID 9328850
- [Background] Bruder N, Pellissier D, Grillot P, Gouin F. Cerebral hyperemia during recovery from general anesthesia in neurosurgical patients. Anesth Analg. 2002 Mar;94(3):650-4; table of contents. doi: 10.1097/00000539-200203000-00031. PMID 11867391
- [Background] Rijbroek A, Boellaard R, Vriens EM, Lammertsma AA, Rauwerda JA. Comparison of transcranial Doppler ultrasonography and positron emission tomography using a three-dimensional template of the middle cerebral artery. Neurol Res. 2009 Feb;31(1):52-9. doi: 10.1179/174313208X325191. Epub 2008 Jul 25. PMID 18662500
- [Background] Sorond FA, Hollenberg NK, Panych LP, Fisher ND. Brain blood flow and velocity: correlations between magnetic resonance imaging and transcranial Doppler sonography. J Ultrasound Med. 2010 Jul;29(7):1017-22. doi: 10.7863/jum.2010.29.7.1017. PMID 20587424
- [Background] Macmillan CS, Andrews PJ. Cerebrovenous oxygen saturation monitoring: practical considerations and clinical relevance. Intensive Care Med. 2000 Aug;26(8):1028-36. doi: 10.1007/s001340051315. PMID 11030158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 11.01.2012-01.31.2013 Study location: Huashan Hospital Fudan University Location Type: Medical centre affiliated to medical university
Pre-assignment Details: Transcranial doppler (TCD) and head CT-scan was used to exclude patients with intracranial hypertension,cerebrovascular diseases, or metastatic brain tumor.
Groups:
- Craniotomy Group: Patients who are scheduled for selective supratentorial tumor removal surgery will be randomly chosen and recruited.
  Transcranial Doppler (TCD) measures,jugular venous bulb catheterization, radial artery catheterization, and tumor removal surgery under general anesthesia will be performed.
- Abdominal Surgery Group: Randomly chosen patients undergoing selective abdominal surgery. Transcranial Doppler measures,radial artery catheterization, and abdominal surgery under general anesthesia will be performed.
Period: Overall Study
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdominal Surgery Group | Craniotomy Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.6 (8.2) | 47.3 (7.6) | 47.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 16 | 17 | 33
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60
Duration of Surgery [Mean (Standard Deviation); unit: minute] | 207 (49) | 214 (38) | 211 (43)

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Flow Velocity in Middle Cerebral Artery
Description: It was the baseline mean blood flow velocity in middle cerebral artery.
Time Frame: before general anesthesia
Population: The number of participants for analysis was determined by sample estimation equation of cohort study. In the equation, the hyperemia frequency from literature and pre-study was used.
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 30
cm/s | 63.7 (6.7) | 61.8 (8.1)
Statistical Analysis 1: Comparison: Craniotomy Group vs Abdominal Surgery Group; H0: Mean Blood Flow Velocity in Middle Cerebral Artery of the 2 groups are the same before anesthesia. Power calculation: beta=0.2, alpha=0.05, two-tailed; Test type: Superiority or Other; p = 0.554, Wilcoxon (Mann-Whitney) — Bonferroni correction is used when P-value is significant

2. Primary Outcome: Mean Blood Flow Velocity in Middle Cerebral Artery
Time Frame: after surgery at extubation (average surgery duration: craniotomy group 214min, abdominal group 207min)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 30
cm/s | 95.7 (16.9) | 63.6 (7.7)
Statistical Analysis 1: Comparison: Craniotomy Group vs Abdominal Surgery Group; H0: Mean Blood Flow Velocity in Middle Cerebral Artery of the 2 groups are the same at extubation. Power calculation: beta=0.2, alpha=0.05, two-tailed; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Bonferroni correction is used when P-value is significant

3. Primary Outcome: Mean Blood Flow Velocity in Middle Cerebral Artery
Time Frame: 30min after extubation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 30
cm/s | 82.5 (12.0) | 62.0 (8.0)
Statistical Analysis 1: Comparison: Craniotomy Group vs Abdominal Surgery Group; H0: mean blood flow velocity in middle cerebral artery of the 2 groups are the same 30min after extubation. Power calculation: beta=0.2, alpha=0.05, two-tailed; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Bonferroni correction is used when P-value is significant

4. Primary Outcome: Mean Blood Flow Velocity in Middle Cerebral Artery
Time Frame: 60min after extubation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 30
cm/s | 77.0 (12.1) | 61.2 (7.9)
Statistical Analysis 1: Comparison: Craniotomy Group vs Abdominal Surgery Group; H0: mean blood flow velocity in middle cerebral artery of the 2 groups are the same 60min after extubation. Power calculation: beta=0.2, alpha=0.05, two-tailed; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Bonferroni correction is used when P-value is significant

5. Primary Outcome: Mean Blood Flow Velocity in Middle Cerebral Artery
Time Frame: 90min after extubation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 30
cm/s | 72.8 (11.0) | 60.1 (8.0)
Statistical Analysis 1: Comparison: Craniotomy Group vs Abdominal Surgery Group; H0: mean blood flow velocity in middle cerebral artery of the 2 groups are the same 90min after extubation. Power calculation: beta=0.2, alpha=0.05, two-tailed; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Bonferroni correction is used when P-value is significant

6. Primary Outcome: Mean Blood Flow Velocity in Middle Cerebral Artery
Time Frame: 120min after extubation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 30
cm/s | 69.7 (9.0) | 59.2 (7.8)
Statistical Analysis 1: Comparison: Craniotomy Group vs Abdominal Surgery Group; H0: mean blood flow velocity in middle cerebral artery of the 2 groups are the same 120min after extubation. Power calculation: beta=0.2, alpha=0.05, two-tailed; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Bonferroni correction is used when P-value is significant

7. Primary Outcome: Oxygen Saturation of Jugular Venous Bulb
Time Frame: before general anesthesia
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 0
percentage of oxygen saturation | 60.9 (3.7) |

8. Primary Outcome: Oxygen Saturation of Jugular Venous Bulb
Time Frame: at extubation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 0
percentage of oxygen saturation | 81.4 (7.4) |

9. Primary Outcome: Oxygen Saturation of Jugular Venous Bulb
Time Frame: 30min after extubation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 0
percentage of oxygen saturation | 77.0 (6.4) |

10. Primary Outcome: Oxygen Saturation of Jugular Venous Bulb
Time Frame: 60min after extubation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 0
percentage of oxygen saturation | 71.8 (6.5) |

11. Primary Outcome: Oxygen Saturation of Jugular Venous Bulb
Time Frame: 90min after extubation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 0
percentage of oxygen saturation | 68.8 (6.4) |

12. Primary Outcome: Oxygen Saturation of Jugular Venous Bulb
Time Frame: 120min after extubation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Craniotomy Group | Abdominal Surgery Group
Number analyzed (Participants) | 30 | 0
percentage of oxygen saturation | 66.9 (5.9) |

ADVERSE EVENTS:
Groups:
- Craniotomy Group: Randomly chosen patients undergoing selective craniotomy surgery. Transcranial Doppler measures,jugular venous bulb catheterization, radial artery catheterization, and craniotomy under general anesthesia will be performed.
Arm/Group | Abdominal Surgery Group | Craniotomy Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
The study population was not homogenous according to tumor size and location.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes